CLINICAL TRIAL: NCT01890304
Title: Diffusion Tensor Imaging (DTI) Compared to Serum Biomarkers and Standard Clinical Measures of Concussion in Female and Male Collegiate Athletes: a Longitudinal Survey Across the College Years.
Brief Title: Longitudinal Study of Traumatic Brain Injury (TBI) in (University of Florida) UF Athletes
Acronym: GATOR TBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Available MRI scan unable to collect required data elements.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68-2013
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; Concussion; Sports related injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Resonance Imaging (MRI) (Other): Athletes at risk for mild traumatic brain injury during the course of competitive play or practice. An MRI will be obtained at study entry, following any TBI occuring during sanctioned practice or play, and at study exit.
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — MRI will be obtained at study entry, following any TBI occuring during sanctioned practice or play, and at study exit.

SUMMARY:
To identify the changes in the brain following repeated sports-related concussion in men's football, women's soccer, and women's lacrosse college athletes by reviewing the findings of MRI studies that look at the structure of the brain and the appearance of the white matter at baseline, during the acute phase of a concussive injury, and upon completion of collegiate athletic play and correlate these findings with standard clinical measures.

DETAILED DESCRIPTION:
This proposal seeks to study Diffusion Tensor Imaging and functional MRI of the brain at 1) baseline, 2) after concussion and 3) at the end of an athlete's college career. Findings will be compared to standard clinical measures already performed in the management of concussion at the University of Florida Athletic Association and to serum biomarkers already being obtained as part of a UF/ Banyan Biomarker Study. As in the biomarker study, UF athletes on teams with higher incidences of sports related concussion; men's football, women's soccer, and women's lacrosse will be offered enrollment.

Longitudinal examinations will allow identification and quantification of concussive DTI findings as comparisons can be made to the individual athlete's baseline data. This will provide valuable correlation of imaging findings with severity of clinical symptoms at the time of injury and also with timing of return to play.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and active UF student athlete in Mens Football, Womens Soccer, or Womens Lacrosse.
* Age 18-30

Exclusion Criteria:

* Contraindications to MRI, such as retained metal
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Fractional Anisotropy (FA) | Change in baseline up to 5 years.
  Changes in FA values will assessed in the white matter of the brain at the time points noted.

SECONDARY OUTCOMES:
Neuropsychometric testing | Change in baseline up to 5 years.
  Correlation of standard neuropsychometric testing will be compared with results of MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Peters, MD, Principal Investigator — Associate Professor of Radiology
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States